CLINICAL TRIAL: NCT03765866
Title: Viscoelastic Guided Goal Directed Resuscitation of Severely Injured Patients
Brief Title: Rotational Thromboelastometry Activated Transfusion In Trauma Trial
Acronym: ROTATE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 022015-093
Record Dates: First submitted 2016-05-23; First posted 2018-12-05 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Trauma
Keywords: rotational thromboelastometry; viscoelastic test; coagulopathy; trauma; hemorrhage
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massive Transfusion Protocol Guided (No Intervention): Clinicians will only transfuse patients according to standard massive transfusion protocol (MTP)
- Thromboelastometry guided transfusion (Experimental): Clinicians will transfuse patients according to ROTEM results.
  Interventions: Procedure: Thromboelastometry guided transfusion

INTERVENTIONS:
Procedure: Thromboelastometry guided transfusion — Comparing resuscitation strategies with standard MTP v.s. ROTEM guided MTP
  Arms: Thromboelastometry guided transfusion

SUMMARY:
This is a randomized controlled trial to compare viscoelastic (VE) guided resuscitation to fixed-ratio resuscitation in trauma patients with hemorrhagic shock on the utilization of blood products, effects on coagulation and inflammatory mediators, and how these strategies affect post resuscitation adverse events.

DETAILED DESCRIPTION:
This is an open labeled study as the VE guided resuscitation will be based on the visible VE results. Aim 1 will compare the number of blood products utilized in each resuscitation strategy. Aim 2 will analyze the coagulation and inflammatory mediators in each resuscitation strategy to determine if there is a difference in the mechanism of coagulopathy. Aim 3 will determine if the different resuscitation strategies have an effect on post resuscitation adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Trauma patient
2. MTP Activation
3. Only patients ≥ 14 years old
4. Alive at 31 mins after arrival in ED

Exclusion Criteria:

1. Transfer from OSH
2. Received CPR for more than 5 mins
3. Burned
4. Pregnant or Prisoner
5. Known DNR
6. Jehovah's witness

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Change in number of blood products utilized at 24 hours | 24 hours from time of randomization
  Number of blood products utilized during that time frame will be recorded to determine if change in resuscitation strategies result in measurable differences

SECONDARY OUTCOMES:
Change in coagulation profile | 0 hours and 30 days
  Analyze coagulation profiles in each resuscitation strategy to determine if there is a change in the mechanism of coagulopathy
Change in inflammatory mediators | 0 hours and 30 days
  Analyze inflammatory mediators in each resuscitation strategy to determine if there is a change in the mechanism of coagulopathy
Changes in Resuscitation strategy-related adverse events | 30 days after admission
  Rate of resuscitation strategies-related adverse events as a composite, including (transfusion related acute lung injury, transfusion associated circulatory overload, hyperkalemia, hypocalcemia, allergic reaction, hemolysis and transfusion transmitted infection)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Cripps, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] Schlimp CJ, Voelckel W, Inaba K, Maegele M, Schochl H. Impact of fibrinogen concentrate alone or with prothrombin complex concentrate (+/- fresh frozen plasma) on plasma fibrinogen level and fibrin-based clot strength (FIBTEM) in major trauma: a retrospective study. Scand J Trauma Resusc Emerg Med. 2013 Oct 8;21:74. doi: 10.1186/1757-7241-21-74. PMID 24103457